CLINICAL TRIAL: NCT00400998
Title: A Randomised, Double Blind, Placebo Controlled, 2-way Crossover, 3 Phase Study, to Investigate the Trial Models, Vienna Challenge Chamber, in and Out of Season, and Park Study in Season and the Clinical Efficacy of Rpt Doses of Fluticasone Propionate in Subjects With Seasonal Allergic Rhinitis
Brief Title: Investigate Two Trial Models; Vienna Challenge Chamber (in and Out of Season) and Park Study (in Season) Using a Drug for Seasonal Allergic Rhinitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Research Consult GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: HH3104994
Record Dates: First submitted 2006-11-15; First posted 2006-11-17 (Estimated); Last update posted 2018-01-10 (Actual); Status verified 2018-01

CONDITIONS: Allergic Rhinitis; Rhinitis, Allergic, Seasonal
Keywords: Seasonal Allergic Rhinitis; Quality of Life; Efficacy; Validation; Fluticasone Propionate
MeSH Terms: conditions — Rhinitis, Allergic; Rhinitis, Allergic, Seasonal | interventions — Fluticasone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Vienna Challenge Chamber in season (Phase 3) (Placebo Comparator): Phase 3 will consist of two treatment periods each lasting 8 days, with a 10 day wash-out between each treatment period.
  Subjects will administer 200micrograms (μg) fluticasone propionate or fluticasone propionate matched placebo nasal spray, once daily for 8 days. Dosing will be supervised on the first and last days of each treatment period (Day 1 and Day 8).
  Immediately following the last dose received on Day 8 the subject's signs and symptoms will be monitored: subjective symptom score every 15 minutes for rhinomanometry and measurement of nasal secretion every 30 minutes, and FEV1, AEs and symptoms of local irritancy.
  Interventions: Drug: Fluticasone Propionate; Other: Matched FPANS placebo
- Vienna Challenge Chamber out of season (Phase 1) (Placebo Comparator): Phase 1 will consist of two treatment periods each lasting 8 days, with a 10 day wash-out between each treatment period.
  Subjects will administer 200μg fluticasone propionate or fluticasone propionate matched placebo nasal spray, once daily for 8 days. Dosing will be supervised on the first and last days of each treatment period (Day 1 and Day 8).
  Immediately following the last dose received on Day 8 the subject's signs and symptoms will be monitored: subjective symptom score every 15 minutes for rhinomanometry and measurement of nasal secretion every 30 minutes, and FEV1, AEs and symptoms of local irritancy.
  An intermediate study follow-up visit will take place 7-14 days after the last dose is received in treatment period 2.
  Interventions: Drug: Fluticasone Propionate; Other: Matched FPANS placebo
- Park In Season (Phase 2) (Placebo Comparator): Phase 2 will consist of 2 treatment periods lasting either 8 to 14 days (D) (depending on out-door conditions). There will be a 10D wash-out between this treatment period in Phase 2 and that in Phase 3.
  Subjects will administer 200μg fluticasone propionate (or fluticasone propionate matched placebo nasal spray, once daily up to 14D, with dosing supervised on the first and last days of each treatment period (D1 and either D8 or up to D14).
  Immediately following the last dose received on either D8 or up to D14 baseline measures will be taken (time = 0). The subject is then taken by bus to the Park and the first measurement will be taken 15 minutes after the subjects leave the bus and enter the Park.
  Immediately following the last dose received on D8 or up to D14 the subject's signs and symptoms will be monitored: subjective symptom score every 15 minutes for rhinomanometry and measurement of nasal secretion every 30 minutes, and FEV1, AEs and symptoms of local irritancy
  Interventions: Drug: Fluticasone Propionate; Other: Matched FPANS placebo

INTERVENTIONS:
Drug: Fluticasone Propionate — Subjects will receive the following treatment regimen over one of two dosing periods within each of the three study phases:
  - Intranasal FPANS (Fluticasone Propionate aqueous nasal spray) 200 mcg once daily for 8 to 14 days i.e. 4 actuations (2 per nostril) daily, where each actuation delivers a volume of 100 mcL (microlitres) i.e. 50 mcg fluticasone propionate.
Other: Matched FPANS placebo — Subjects will receive the following placebo treatment regimen over one of two dosing periods within each of the three study phases:
  * Intranasal FPANS placebo once daily for 8 to 14 days (i.e. 4 actuations (2 per nostril) daily, where each actuation delivers a volume of 100 mcL.

SUMMARY:
The aim of the study is to investigate the trial models, Vienna Challenge Chamber (VCC), in and out of season, and Park Study in season and the clinical efficacy of repeat doses of fluticasone propionate in subjects with seasonal allergic rhinitis.

DETAILED DESCRIPTION:
The aim of the study is to investigate the trial models, Vienna Challenge Chamber (VCC), in and out of season, and Park Study in season and the clinical efficacy of repeat doses of fluticasone propionate in subjects with seasonal allergic rhinitis. This will be a single-centre, randomised, double-blind, placebo-controlled, 3 phase study in 40 male or female subjects with seasonal allergic rhinitis. The subjects will be randomised to receive either fluticasone propionate aqueous nasal spray or matched placebo. The study consists of three phases with each phase consists of 2 treatment periods. A screening visit will be followed by Phase 1 (Vienna Chamber Challenge out of season), Phase 2 (Park Study, in season) and Phase 3 (Vienna Chamber Challenge in season). There will be a follow-up visit after Phase 1 and Phase 2 & 3 will be separated by a 10 day wash-out period. A follow-up visit will be completed 7-14 days after the last received dose. Intranasal fluticasone propionate will be administered daily for 8 days in the VCC and up to 14 days in the Park Study. Primary assessment will consist of major symptoms complex (MSC) during a 5-hour pollen allergen challenge in the Vienna Challenge Chamber (VCC) following final dosing on Day 8 and following final dosing between Day 8 and Day 14 in the Park Study. In addition, nasal flow measured by anterior rhinomanometry, wet tissue weight (as a surrogate of nasal secretion) and categorical scores for ocular symptoms, cough, itchy throat and itchy ears will be measured on day 8 (VCC) or on a day between 8-14 (Park).

ELIGIBILITY:
Inclusion Criteria:

* The subject is healthy. Healthy subjects are defined as individuals who are free from clinically significant illness or disease as determined by their medical history (including family), physical examination, laboratory studies, and other tests.
* They have a history of seasonal allergic rhinitis
* Exhibit a moderate response to 1500 grass pollen grains per cubic metre after 2 hours in the Vienna Challenge Chamber at screening or within 12 months preceding the screening visit. A moderate response is defined as a total nasal symptom score of at least 6. (Total nasal symptom score is the sum of obstruction, rhinorrhoea, itch and sneeze, each of which has been scored on a scale from 0 to 3).
* They have a positive skin prick test (wheal size equal to or more than 4mm) for grass pollen at or within the 12 months preceding the screening visit.
* They have a positive RadioAllergoSorbent Test (RAST) (equal to or more than class 2) for grass pollen at or within the 12 months preceding the screening visit.
* They have demonstrated an ability to use the intranasal spray
* There are no conditions or factors which would make the subject unlikely to be able to stay in the chamber for 5 hours.
* They are capable of giving informed consent which includes compliance with the requirements and restrictions listed in the consent form
* They are available to complete all study measurements

Exclusion Criteria:

* Pregnant or nursing females.
* Female subjects of childbearing potential who are unwilling or unable to use an appropriate method of contraception [i.e. implants of levonorgestrel, injectable progesterone, an acceptable intra-uterine device (IUD) (any IUD with a failure rate of less than 1% per year), oral contraceptives or any other method with a failure rate of <1% per year] for at least two weeks prior to the first dose of study medication and should continue using the same contraceptive measure until the final pregnancy test has been performed (not less than 72 hours after treatment). Alternatively they may be surgically sterilised (refer to section 6.4) or remain abstinent for 2 weeks before exposure to study drug.
* On examination the subject is found to have any structural nasal abnormalities or nasal polyposis, a history of frequent nosebleeds, recent nasal surgery or recent (within 3 weeks) or ongoing upper respiratory tract infection which in the responsible physician's opinion renders the subject unsuitable for participation in the study
* The subject has any respiratory disease other than mild stable asthma that is controlled with occasional use of as-needed short-acting beta-agonists and associated with normal lung function.
* The subject is likely to be unable to abstain from salbutamol use for 8 hours before a challenge
* The subject has a history of drug or other allergy that, in the opinion of the responsible physician, contraindicates their participation.
* The subject has participated in a study with a new molecular entity during the previous 3 months or in any clinical study in the previous 2 months
* The subject is concurrently participating in another clinical study in which the subject is or will be exposed to an investigational or a non-investigational drug or device.
* The subject is currently taking regular (or a course of) medication whether prescribed or not, including steroids, vitamins and herbal remedies (e.g. St. John's Wort). Paracetamol and occasional as needed use of short-acting beta agonists is permitted
* The subject regularly, or on average, drinks more than 3 units of alcohol per day - where 1 unit = ½ pint of beer (284milliliteres mL), or 1 glass of wine (125mL), or 1 measure of spirit (25mL).
* The subject is at risk of non-compliance with the study procedures/restrictions.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 41 (Actual)
Dates: Start 2006-03; Primary Completion 2006-11 (Actual); Study Completion 2006-11 (Actual)

PRIMARY OUTCOMES:
Weighted mean major symptom complex (MSC) sneeze, nasal itch, rhinorrhoea and itching eyes following 5 hours spent in the Vienna Challenge Chamber (VCC), in and out of season, and 5 hours in the Park Study in season. | 0-5 hour after last dose in either model

SECONDARY OUTCOMES:
Weighted Mean Total Nasal Symptom Score (TNSS) in both in-Chamber and Park studies | 0-5 hour after last dose in either model
Weighted mean eye symptom score in both in-Chamber and Park studies | 0-5 hour after last dose in either model
Weighted mean global symptom score in both in-Chamber and Park studies | 0-5 hour after last dose in either model
Weighted mean nasal airflow resistance in both in-Chamber and Park studies | 0-5 hour after last dose in either model
Mean nasal secretion weight in both in-Chamber and Park studies | 0-5 hour after last dose in either model
Forced Expiratory Volume in 1 second (FEV1) in both in-Chamber and Park studies | 0-5 hour after last dose in either model
Adverse Events in both in-Chamber and Park studies | 0-5 hour after last dose in either model
Symptoms of local irritancy in both in-Chamber and Park studies | 0-5 hour after last dose in either model
Quality of life in both in-Chamber and Park studies | 0-5 hour after last dose in either model
Time until a 20% reduction is seen in TNSS, mean and global symptom scores, Nasal airflow resistance, Nasal secretion weight and FEV1 | 2 hour after last dose in either model

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Vienna, Austria